CLINICAL TRIAL: NCT02827123
Title: A Comparison of McGrath MAC Videolaryngoscopy and Macintosh Laryngoscopy for Orotracheal Intubation in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Ji Eun Kim, Assitant professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AJIRB-MED-DE4-16-150
Record Dates: First submitted 2016-07-03; First posted 2016-07-11 (Estimated); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Anesthesia, Endotracheal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Mcgrath group (Experimental): Orotracheal intubation with McGrath MAC videolaryngoscopy
  Interventions: Device: McGrath MAC videolaryngoscopy
- Macintosh group (Placebo Comparator): Orotracheal intubation with Macintosh laryngoscopy
  Interventions: Drug: Macintosh Laryngoscopy

INTERVENTIONS:
Device: McGrath MAC videolaryngoscopy — Orotracheal intubation with McGrath MAC videolaryngoscopy after anesthetic induction
  Arms: Mcgrath group
Drug: Macintosh Laryngoscopy — Orotracheal intubation with Macintosh Laryngoscopy after anesthetic induction
  Arms: Macintosh group

SUMMARY:
The primary purpose of this study is to investigate the effects of McGrath MAC videolaryngoscopy on the intubation time for orotracheal intubation in children.

The secondary purpose of this study is to investigate the effects of McGrath MAC videolaryngoscopy on Cormack and Lehane Grade for orotracheal intubation in children.

ELIGIBILITY:
Inclusion Criteria:

* orotracheal intubation under general anesthesia

Exclusion Criteria:

* oral lesions, congenital anomaly, cervical spine instability, rapid sequence intubation

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2016-07; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Intubation time | through intubation completion, an average of 30 second
  Time interval between laryngoscopy passing the teeth to the confirming of end tidal CO2

SECONDARY OUTCOMES:
The degree of glottic exposure as assessed by Cormack and Lehane Grade | Up to 5 second after laryngoscopy passing the teeth
  Grade 1: full view of glottis, grade 2: Partial view of glottis, grade 3:only epiglottis seen, grade 4:neither glottis nor epiglottis seen

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Ajou University School of Medicine, Suwon, Seoum, South Korea